CLINICAL TRIAL: NCT06041659
Title: Functional Magnetic Resonance-Based Observations of Brain Networks and Cerebrovascular Reactivity in Patients With Moyamoya Disease Under Anesthetic Sedation, A Prospective Observational Cohort Study
Brief Title: Functional Magnetic Resonance-Based Observations of Brain Networks in Moyamoya Disease Patients Under Anesthesia
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yuming Peng, Clinical Professor, Beijing Tiantan Hospital
Other Study IDs: 2023022
Record Dates: First submitted 2023-09-11; First posted 2023-09-18 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Moyamoya Disease
Keywords: Moyamoya Disease; Cerebral Network; Cognitive Function; Anesthesia
MeSH Terms: conditions — Moyamoya Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Moyamoya disease is characterized by progressive stenosis of the genesis of the distal internal carotid arteries bilaterally and progressive generation of compensatory pathological vascular networks at the basis cranii, and these pathological vasculature has poor vascular reactivity. Perioperative circulatory management of patients with smoky vessels to ensure perfusion of brain tissue and integrity of brain network during surgery to minimize postoperative impairment of neurological functions, including motor, sensory, emotional and cognitive functions, is the key point of perioperative circulatory management of moyamoya disease. Functional Magnetic Resonance Imaging (fMRI) has been routinely used in various cerebrovascular diseases to further evaluate cerebrovascular reserve and cerebral network connectivity. The purpose of this study is to observe the changes in cerebral blood flow, cerebral oxygen metabolism, cerebral oxygen metabolism rate, and cerebral network connectivity in adult patients with moyamoya disease in cerebral ischemia-sensitive areas under anesthesia to provide a basis for exploring anesthesia management to improve cognitive function and cerebral network connectivity in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moyamoya disease scheduled for direct or indirect intracranial and extracranial revascularization surgery
* Age between 18-65 years
* Obtain written informed consent.

Exclusion Criteria:

* Patients with preoperative claustrophobia, sensory or motor aphasia that are unable to understand and cooperate with the examination
* Preoperative cranial imaging suggesting cerebral infarction lesion diameter >15mm
* Patients allergic to anesthetic drugs
* Metal implants in the body
* Undergoing other experimental drug or instrumentation trials

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We plan to recruit consecutive patients with moyamoya disease who are to undergo direct or indirect revascularization surgery from August 2023 to December 2025 at Beijing Tiantan Hospital of Capital Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of brain functional network | Before sedation, after sedation and after maintenan the blood pressure at baseline 100%-120% for 15min

SECONDARY OUTCOMES:
Postoperative delirium | Day1-5 after surgery
Electroencephalogram changes | Before sedation, after sedation and after maintenan the blood pressure at baseline 100%-120% for 15min

CONTACTS AND LOCATIONS:
Overall Officials: Shu Li, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided